CLINICAL TRIAL: NCT04377789
Title: The Possible Effect of Quercetin on Prophylaxis and Treatment of COVID-19
Brief Title: Effect of Quercetin on Prophylaxis and Treatment of COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Collaborators: Orbiteratec (funding) (Unknown)
Responsible Party: Principal Investigator, Hasan Onal, Professor, Kanuni Sultan Suleyman Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KSSEAH--0058
Record Dates: First submitted 2020-05-01; First posted 2020-05-06 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- non-quercetin group (No Intervention): Participants, who accept to enroll the study without having quercetin prophylaxis and who do not have a history of COVID-19, will be in this group.
- quercetin prophylaxis group (Active Comparator): Participants, who takes a daily dose of 500mg quercetin and who not have a history of COVID-19, will be in this group.
  Interventions: Dietary Supplement: Quercetin Prophylaxis
- quercetin treatment group (Active Comparator): Participants, who takes a daily dose of 1000mg quercetin and who are proven cases for COVID-19, will be in this group.
  Interventions: Dietary Supplement: Quercetin Treatment

INTERVENTIONS:
Dietary Supplement: Quercetin Prophylaxis — a daily dose of quercetin (500mg) will be taken by non-COVID-19 intervention group 1
  Arms: quercetin prophylaxis group
Dietary Supplement: Quercetin Treatment — a daily dose of quercetin (1000mg) will be taken by proven COVID-19 cases intervention group 2
  Arms: quercetin treatment group

SUMMARY:
Novel Coronavirus is defined to be the cause of COVID-19, recently. It's known that COVID-19 goes with excessive immune reaction of human body in severe cases. The investigators hypothesize that quercetin, as a strong scavenger and anti-inflammatory agent, can be effective on both prophylaxis and treatment of COVID-19 cases. Therefore, the aim of this study to evaluate the possible role of quercetin on prophylaxis and treatment of COVID-19.

DETAILED DESCRIPTION:
Novel Coronavirus is defined to be the cause of COVID-19, recently. It's known that COVID-19 goes with excessive immune reaction of human body in severe cases. Quercetin is reported to be effective on treatment and prophylaxis of other SARS like coronavirus infections, as a strong antioxidant and scavenger flavonoid without any adverse events. Upon this data, the investigators hypothesize that quercetin can be effective on both prophylaxis and treatment of COVID-19 cases. Therefore, the aim of this study to evaluate the possible role of quercetin on prophylaxis and treatment of COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* moderate-high risk for COVID-19
* obtained informed consent

Exclusion Criteria:

* declined to participate
* genetic/chromosomal abnormalities
* any kind of sensitivity or allergy for quercetin
* history of previous hypersensitivity with quercetin

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 447 (Actual)
Dates: Start 2020-03-20 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of COVID-19 calculated using a questionnaire | 3 months
  Prevalence of COVID-19 in prophylaxis and sham group will be calculated using a questionnaire including hospital records
Standardized Mortality rate | 3 months
  Mortality rate will be compared between two groups

SECONDARY OUTCOMES:
Morbidity rate | 3 months
  Morbidity rates besides recovery rates from COVID-19 will be documented

CONTACTS AND LOCATIONS:
Locations (1):
- Kanuni Sultan Suleyman Training and Research Hospital, Istanbul, Turkey (Türkiye)